CLINICAL TRIAL: NCT03461536
Title: Ultrasound First Clinical Decision Support for Suspected Nephrolithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 18-24325
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, investigators, and outcome assessors will be blinded to study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Decision Support (Active Comparator): Participants in this arm will receive the study intervention, the clinical decision support.
  Interventions: Behavioral: Ultrasound-first Clinical Decision Support tool
- Usual care (No Intervention): Participants in this arm will not receive the the clinical decision support tool.

INTERVENTIONS:
Behavioral: Ultrasound-first Clinical Decision Support tool — Intervention: The intervention is the CDS tool, which consists of 4 components:
  1. Four questions which assess the appropriateness of ultrasound for this patient
  2. A link to the evidence
  3. Buttons to remove CT scan and order ultrasound
  4. If the CT scan order is kept, reasons why ultrasonography is not appropriate The CDS tool will be placed or integrated into EPIC, at the point of order entry. The tool will be triggered by an order for CT scan for kidney stone.
  Appropriateness criteria for ultrasound:
  1. Adults aged >18 and < 76
  2. Non-obese (men < 285lbs, women < 250lbs)
  3. Low risk of Stone Emergency (Obstructing stone and any of the following: urosepsis, renal deterioration, post kidney transplant, solitary kidney, intractable symptoms)
  4. Low risk of clinically significant alternative diagnosis (e.g. appendicitis, cholecystitis, AAA, ovarian torsion) If all responses are affirmative, then the subject should receive US, and US order is provided.
  Arms: Clinical Decision Support

SUMMARY:
This is a randomized trial to determine the effectiveness of a clinical decision support tool on image ordering for patients with suspected nephrolithiasis. Patients who present with acute unilateral flank or abdominal pain in whom emergency department providers suspect nephrolithiasis will receive either the clinical decision support tool or no tool (usual care).

DETAILED DESCRIPTION:
CT scan is overused for patients who present to the ED with suspected nephrolithiasis (acute flank or abdominal pain). The investigators have developed a clinical decision support (CDS) tool to identify those patients in whom ultrasound is appropriate. The CDS tool is based on the Study of Ultrasonography vs. Computed Tomography for Suspected Nephrolithiasis in the Emergency Department.

The goal of this study is to assess the effectiveness of a clinical decision support (CDS) tool to improve advanced imaging for suspected nephrolithiasis in the ED. The investigators hypothesize those randomized to receiving the CDS tool will receive CT less often (and less radiation) compared to those receiving control. Also, the investigators hypothesize those randomized to receiving CDS will have a similar ED length of stay and rate of unexpected ED return as those receiving control.

Study design: Randomized trial of a CDS tool embedded in the electronic health record for patients with suspected nephrolithiasis. The study will be conducted at UCSF Department of Emergency Medicine.

Study subjects: The investigators will enroll adult patients who present to the UCSF ED who present with "suspected nephrolithiasis", which is defined as those with symptoms of nephrolithiasis for whom an ED provider orders a CT scan for suspected nephrolithiasis. Symptoms of nephrolithiasis include acute unilateral flank and/or abdominal pain, typically described as severe and colicky. The pain is accompanied by nausea, vomiting, and urinary symptoms, such as hematuria. The CT imaging studies emergency physicians typically order for suspected nephrolithiasis include CT scan without contrast; however a substantial minority of patients receive CT scan with contrast, and CT scan with and without contrast for acute flank pain, suspected nephrolithiasis.

Sampling, recruiting and retaining subjects: The investigators will enroll consecutive patients who present to the ED with the selection criteria. Those with suspected nephrolithiasis but have an exclusion criteria will be recorded and compared to those who were enrolled. Eligible patients will be randomized to either receiving CDS recommendations or no CDS recommendations. Subjects will not receive informed consent, and will not be contacted by staff.

Intervention: The intervention is the CDS tool, which consists of 4 components:

1. Four questions which assess the appropriateness of ultrasound for this patient
2. A link to the evidence
3. Buttons to remove CT scan and order ultrasound
4. If the CT scan order is kept, reasons why ultrasonography is not appropriate

The CDS tool will be placed or integrated into EPIC, at the point of order entry. The tool will be triggered by an order for CT to identify or rule out kidney stone.

Co-primary outcomes: Proportion of study arm who receive CT, and radiation dose. Proportion of study arm who receive CT is defined as #CT scans ordered/#patients in study arm. Radiation dose will be reported as median radiation dose in mSv. The secondary outcomes will include proportion of patients with an unscheduled return due to missed diagnosis, cost, ED length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who present to the ED with flank or abdominal pain for whom ED provider orders a CT scan for suspected nephrolithiasis

Exclusion Criteria:

- Previous enrollment into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
CT use | During the index emergency department visit
  Whether the patient received CT scan
Radiation Dose | During the index emergency department visit
  Radiation dose in millisieverts

SECONDARY OUTCOMES:
Return Visit | Within 1 week of the ED index visit
  Return visits to ED with hospitalization
ED Length of Stay | During the index emergency department visit
  ED Length of Stay
Cost | During the index emergency department visit
  Total cost

CONTACTS AND LOCATIONS:
Overall Officials: Ralph C Wang, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang RC, Fahimi J, Dillon D, Shyy W, Mongan J, McCulloch C, Smith-Bindman R. Effect of an ultrasound-first clinical decision tool in emergency department patients with suspected nephrolithiasis: A randomized trial. Am J Emerg Med. 2022 Oct;60:164-170. doi: 10.1016/j.ajem.2022.08.015. Epub 2022 Aug 10. PMID 35986979